CLINICAL TRIAL: NCT01576679
Title: A Double Blind, Randomized Controlled Trial Examining the Efficacy of the Use of Tissue Plasminogen Activator (tPA) in Intra-abdominal Collections in Children - a Prospective Study
Brief Title: Safety and Efficacy of the Use of Tissue Plasminogen Activator (tPA) in Intra-Abdominal Collections in Children - A Prospective Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: very slow accrual.
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Bairbre Connolly, Project Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000029136
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Intra-abdominal Abscess
Keywords: intra-abdominal; abscess; tPA; alteplase; cathflo
MeSH Terms: conditions — Abdominal Abscess; Abscess | interventions — Tissue Plasminogen Activator; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tPA (Experimental): tissue Plasminogen Activator
  Interventions: Drug: Cathflo (Alteplase)
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Cathflo (Alteplase)
  Arms: tPA
Drug: Saline
  Arms: Placebo

SUMMARY:
The objective of this study is to establish the efficacy of tPA when used in pediatric intra-abdominal abscesses immediately after percutaneous drainage, irrespective of the ultrasound appearance or consistency of the drained fluid.

DETAILED DESCRIPTION:
The use of tPA in pediatric abdominal abscesses is poorly defined. The indications are somewhat subjective and the dosage guidelines vary between institutions. Some studies have suggested that it be administered at, or soon after, the time of drainage if the ultrasound appearance of the collection is complex and/or septated, or if the initial aspirated contents are thick and viscous. Both criteria are difficult to accurately define and implement. In many instances, when there is minimal ongoing drainage despite follow-up ultrasound appearances suggesting a significant residual collection, tPA is administered several days following the initial procedure.

The purpose of this study is to establish the efficacy of tPA in the initial treatment of all pediatric intra-abdominal abcesses and a standardized manner in which it can be used. This may eventually lead to a change in practice in the management of this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. All patients under the age of 18 years with intra-abdominal bacterial abscesses requiring percutaneous drain insertion (including transrectal drains).
2. Drain(s) must be inserted within the 23hrs prior to enrollment in the study.
3. The underlying diagnosis of the condition will not affect the enrollment of the patient unless it is detailed within the exclusion criteria (section 4.1.2).
4. Patients and parents must have signed informed consent to participate in the study.

Exclusion Criteria:1.

1. Pancreatic abscess (not bacterial in nature)
2. Known coagulation impairment
3. Known central nervous system tumor or abscesses
4. Arteriovenous malformation
5. Aneurysm or history of central nervous system bleeding
6. Hypersensitivity to tPA
7. Recent administration of an investigational drug (within previous 30 days)
8. Pregnancy
9. Breast-feeding
10. Fulminant hepatic failure
11. Proven fistula (as it will alter the drainage time) or any abscess secondary to Crohn's Disease (because fistula existence cannot be excluded)
12. Necrotizing enterocolitis
13. Children requiring 4 or more drains

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Length of time the drain remains insitu | up to 2 weeks
  The primary outcome is the length of time (in hours) the drain remains insitu.
  For the primary outcome the individual abscess will be the unit of measurement; if there are multiple abscesses (up to a maximum of three) in the one patient each abscess will receive the same treatment. In the case of more than one drain being inserted in a single patient, the length of time that each drain remains in situ will be recorded individually.

SECONDARY OUTCOMES:
Documentation of any adverse event | up to 2 weeks
The length of hospital stay | up to 2 months
Rate of resolution of abscess | up to 2 weeks
Return of clinical parameters to normal | up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bairbre Connolly, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No